CLINICAL TRIAL: NCT04667546
Title: Assessment of the Efficacy on the 5th Day of Antibiotic Therapy for Febrile Urinary Tract Infections Among Children From 3 Months to 18 Years Old
Acronym: PEDIU5
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020/530
Record Dates: First submitted 2020-11-16; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Urinary Tract Infections; Pediatric Disorder
MeSH Terms: conditions — Urinary Tract Infections | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient having urinary tract infection (Other): Patients with a confirmed urinary tract infection in accordance with the GPIP (french Pediatric Infectious Disease Group) definition and inclusion criteria.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Patients or their parents will complete a survey at D2, D5, D10 and D28 to assess the presence or absence of a symptom

SUMMARY:
The main objective is to describe the rate of asymptomatic patients after 5 days of effective antibiotic therapy in an uncomplicated febrile urinary tract infection in children between 3 months and 18 years of age.

DETAILED DESCRIPTION:
This is a non-randomised prospective monocentric pilot study whose main objective is to describe the proportion of asymptomatic patients after 5 days of effective antibiotic therapy in an uncomplicated febrile urinary tract infection, in children between 3 months and 18 years of age. After being informed about the study, all patient meeting inclusion criteria will respond to a survey at D2, D5, D10 and D28 to evaluate the persistence of symptoms to determine the effectiveness of a 5-day course of antibiotic treatment. All patients will be treated in accordance to the French guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Child between 3 months and 18 years old
* Diagnosis of uncomplicated febrile urinary tract infection certain and defined by :

  * Naked fever (without an identifiable source of infection) for at least 24 hours for boys and 48 hours for girls.
  * A urine test strip with at least 2 crosses of leukocyturia ≥ or 1 cross of leukocyturia ≥ with positive nitrituria
  * A cytobacteriological urine test with leukocyturia greater than 10/mm3 in the case of catheterisation or Clean catch or greater than 100/mm3 if the collection is performed by bag (Urinocol®).
  * Positive bacteriological urine culture
  * Response to antibiotic therapy
  * Absence of other diagnoses that could explain the clinical picture

Exclusion Criteria:

* Children under 3 months old
* Immunodepression
* Underlying uropathy or known neurological bladder disease

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of treatment | Day 5
  The main evaluation criteria aims to determine the effectiveness of a 5-day course of antibiotic treatment. Treatment failure is characterised by the presence at Day 5 of clinical signs (abdominal pain, urinary functional signs, urinary burns) and/or a fever ≥ at 38°C and/or a new positive cytobacteriological urine test performed after antibiotic therapy due to the persistence and/or reappearance of symptoms.

SECONDARY OUTCOMES:
Leukocyte count | Day 1
  Leukocyte count (in cell per mm3) in children with uncomplicated febrile urinary tract infections at diagnostic.
Mode of sampling | Day 1
  Leukocyturia rate (cell per mm3), according to the method of collection, on the sample carried out at the first consultation of children with febrile urinary tract infections at diagnostic.
Rate of failure | Day 28
  Measurement of the number of patients presenting a failure at Day 10 or a relapse at 28 days of treatment of a febrile urinary infection. This is characterised by the presence or reappearance of symptoms suggestive of a febrile urinary infection and/or fever without any other possible diagnosis and a positive cytobacteriological urine test with a phenotypically identical micro-organism on the new antibiogram
Procalcitonin levels | Day 1
  Procalcitonin levels (in µg/L) in children with uncomplicated febrile urinary tract infections at diagnostic.
CRP levels | Day 1
  C Reactive Protein (CRP) levels (in mg/l) in children with uncomplicated febrile urinary tract infections at diagnostic.
Polynuclear cell count | Day 1
  Blood polynuclear cell count (in cell per mm3) in children with uncomplicated febrile urinary tract infections at diagnostic.